CLINICAL TRIAL: NCT05487807
Title: Quit4Life+: Adapting and Evaluating a Phone-Based Tobacco Use Cessation Program for People Living With HIV in Uganda and Zambia (Quit4Life+ )
Brief Title: Adapting and Evaluating a Tobacco Use Cessation Program for People Living With HIV in Uganda and Zambia
Acronym: Quit4Life
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Heather Wipfli, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00006; 1U01CA261624 (NIH)
Record Dates: First submitted 2022-07-18; First posted 2022-08-04 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Nicotine Dependence; Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Intervention Model Description: Randomized control trial with 4 arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of Care (No Intervention): This is the baseline group receiving advice to quit.
- Nicotine Replacement (Active Comparator): This group will receive the standard of care and be prescribed nicotine replacement therapy
  Interventions: Drug: Nicotine patch
- Text Messaging (Active Comparator): This group will receive the standard of care and receive text message support
  Interventions: Behavioral: text messaging
- Nicotine replacement and text messaging (Active Comparator): This group will receive the standard of care, be prescribed nicotine replacement therapy, and receive text message support
  Interventions: Drug: Nicotine patch; Behavioral: text messaging

INTERVENTIONS:
Drug: Nicotine patch — Will be receiving nicotine therapy
  Other Names: NicoDerm
  Arms: Nicotine Replacement; Nicotine replacement and text messaging
Behavioral: text messaging — Will be enrolled in an texting app
  Other Names: Text2Quit
  Arms: Nicotine replacement and text messaging; Text Messaging

SUMMARY:
This proposal tests the efficacy of a phone-based tobacco cessation intervention for people living with HIV (PLWH) in comparison to the standard of care (brief advice to quit) and nicotine replacement therapy (nicotine patches) in Uganda and Zambia. This study will provide insight into the efficacy, feasibility, applicability, and affordability of delivering tobacco cessation interventions through health care professionals at HIV treatment centers in two countries with different tobacco use patterns, policy environments, and health care resources. The previously tested SMS-platform to be used in this study is uniquely positioned to be scaled in low- and middle-income countries worldwide, in which case rigorous research showing even modest success in reducing the prevalence of tobacco consumption among PLWH could confer substantial health and economic benefits.

DETAILED DESCRIPTION:
While there is substantial evidence supporting interventions to help tobacco users in the general population quit, little is available relevant to the challenges facing HIV+ tobacco users, especially those living in low-income African countries. This study approaches this gap with the first randomized control trial (RCT) to test the efficacy of a tailored short message service (SMS) based tobacco use cessation intervention on prolonged tobacco use abstinence at 6 months post program initiation in comparison to the standard of care (brief advice to quit) and nicotine replacement therapy (nicotine patches) among PLWH in Uganda and Zambia. This study will provide insight into the efficacy, feasibility, applicability, and affordability of delivering tobacco cessation interventions through health care professionals at HIV treatment centers in two countries with different tobacco use patterns, policy environments, and health care resources and provide needed information to providers and policymakers looking for cost-effective tobacco cessation interventions.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Females who are pregnant, planning to get pregnant, or breastfeeding
* <18 years (underage of consent)
* Visitor, not receiving continuous care at study site
* Not a current daily tobacco user
* Any physical, cognitive, or psychological disabilities that would prevent them from participating in the study
* Illiterate in English and/or local languages
* Does not consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Prolonged tobacco abstinence | 6 months post enrollment
  The primary outcome for this efficacy trial is the proportion of study participants that have prolonged abstinence (i.e., no tobacco use from the target quit date through follow-up) at 3 and 6 months post enrollment measured by self-report and biochemically-verified as recommended by the Society for Research on Nicotine and Tobacco, the biomarker being assessed is urinary cotinine (<12 ng/mL) at 6 months post enrollment

SECONDARY OUTCOMES:
Point Prevalence | 4 weeks, 8 weeks, and 3 months post enrollment
  7 consecutive days of no tobacco use, biochemically-verified at 4 weeks, 8 weeks, and 3 months post enrollment, the biomarker being assessed is urinary cotinine (<12 ng/mL) at 6 months post enrollment, the measurement tool is urine cotinine dip sticks

OTHER OUTCOMES:
Quit attempts | 4 weeks, 8 weeks, and 3 months post enrollment
  Self-reported quit attempts and changes in tobacco use, monitoring survey, health assessment form
Nicotine patch adherence | 4 weeks, 8 weeks, and 3 months post enrollment
  Self-reported adherence to nicotine patch treatment, monitoring survey, health assessment form

CONTACTS AND LOCATIONS:
Locations (2):
- Makerere University, Kampala, Uganda
- University of Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No
Our dissemination strategy will target tobacco and HIV stakeholders including Ministry of Health and other government officials, health care organizations, health facility managers, HIV health care providers, tobacco control professionals, non-governmental organizations engaged in HIV and tobacco control, and PLWH. Our investigators will publish study results through peer-reviewed journals and scientific conferences; generate fact sheets and policy briefs; and disseminate our results through websites, social media, television and radio. We will share the study results in the participating Districts and the Cancer Treatments Centers of America will host a workshop in the final year with regional stakeholders to share the study results and promote tobacco use cessation programming for PLWH throughout Sub-saharan Africa. World Health Organization will assist in disseminating the study findings to other low/middle income countries.

REFERENCES:
- [Background] Lifson AR, Neuhaus J, Arribas JR, van den Berg-Wolf M, Labriola AM, Read TR; INSIGHT SMART Study Group. Smoking-related health risks among persons with HIV in the Strategies for Management of Antiretroviral Therapy clinical trial. Am J Public Health. 2010 Oct;100(10):1896-903. doi: 10.2105/AJPH.2009.188664. Epub 2010 Aug 19. PMID 20724677
- [Background] Jackson-Morris A, Fujiwara PI, Pevzner E. Clearing the smoke around the TB-HIV syndemic: smoking as a critical issue for TB and HIV treatment and care. Int J Tuberc Lung Dis. 2015 Sep;19(9):1003-6. doi: 10.5588/ijtld.14.0813. PMID 26260816
- [Background] Murphy JD, Liu B, Parascandola M. Smoking and HIV in Sub-Saharan Africa: A 25-Country Analysis of the Demographic Health Surveys. Nicotine Tob Res. 2019 Jul 17;21(8):1093-1102. doi: 10.1093/ntr/nty176. PMID 30165688
- [Background] Mitton JA, North CM, Muyanja D, Okello S, Vorechovska D, Kakuhikire B, Tsai AC, Siedner MJ. Smoking cessation after engagement in HIV care in rural Uganda. AIDS Care. 2018 Dec;30(12):1622-1629. doi: 10.1080/09540121.2018.1484070. Epub 2018 Jun 7. PMID 29879856
- [Background] Kruse C, Betancourt J, Ortiz S, Valdes Luna SM, Bamrah IK, Segovia N. Barriers to the Use of Mobile Health in Improving Health Outcomes in Developing Countries: Systematic Review. J Med Internet Res. 2019 Oct 9;21(10):e13263. doi: 10.2196/13263. PMID 31593543
- [Background] Kruse GR, Bangsberg DR, Hahn JA, Haberer JE, Hunt PW, Muzoora C, Bennett JP, Martin JN, Rigotti NA. Tobacco use among adults initiating treatment for HIV infection in rural Uganda. AIDS Behav. 2014 Jul;18(7):1381-9. doi: 10.1007/s10461-014-0737-8. PMID 24638166
- [Result] Hughes JR, Keely JP, Niaura RS, Ossip-Klein DJ, Richmond RL, Swan GE. Measures of abstinence in clinical trials: issues and recommendations. Nicotine Tob Res. 2003 Feb;5(1):13-25. PMID 12745503
- [Result] Baisley K, Baeten JM, Hughes JP, Donnell DJ, Wang J, Hayes R, Watson Jones D, Celum C. Summary measures of adherence using pill counts in two HIV prevention trials: the need for standardisation in reporting. AIDS Behav. 2013 Nov;17(9):3108-19. doi: 10.1007/s10461-013-0542-9. PMID 23801018
- [Result] Schnoll RA, Patterson F, Wileyto EP, Heitjan DF, Shields AE, Asch DA, Lerman C. Effectiveness of extended-duration transdermal nicotine therapy: a randomized trial. Ann Intern Med. 2010 Feb 2;152(3):144-51. doi: 10.7326/0003-4819-152-3-201002020-00005. PMID 20124230
- [Derived] Wipfli H, Arinaitwe J, Goma F, Atuyambe L, Guwatudde D, Phiri MM, Rutebemberwa E, Wabwire-Mangen F, Zulu R, Zyambo C, Guy K, Kusolo R, Mukupa M, Musasizi E, Tucker JS. Usability and cultural adaptation of a text message-based tobacco cessation intervention for people living with HIV in Uganda and Zambia. Addict Sci Clin Pract. 2025 Jul 20;20(1):55. doi: 10.1186/s13722-025-00580-z. PMID 40684230
- [Derived] Guy K, Arinaitwe J, Goma FM, Atuyambe L, Guwatudde D, Zyambo C, Kusolo R, Mukupa M, Musasizi E, Wipfli H. Understanding stigma as a barrier to cancer prevention and treatment: a qualitative study among people living with HIV in Uganda and Zambia. BMJ Open. 2025 Mar 12;15(3):e090817. doi: 10.1136/bmjopen-2024-090817. PMID 40074264
- [Derived] Wipfli H, Arinaitwe J, Goma F, Atuyambe L, Guwatudde D, Phiri MM, Rutebemberwa E, Wabwire-Mangen F, Zulu R, Zyambo C, Guy K, Kusolo R, Mukupa M, Musasizi E, Tucker JS. A phone-based tobacco use cessation program for people living with HIV in Uganda and Zambia: study protocol for a randomized controlled trial. Addict Sci Clin Pract. 2024 Jan 19;19(1):6. doi: 10.1186/s13722-024-00438-w. PMID 38243301